CLINICAL TRIAL: NCT04207216
Title: Use of Alternative Therapy in Psoriasis Vulgaris Patients
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Melek Aslan Kayıran, Spesialist Dermatologist Doctor, Istanbul Medeniyet University
Other Study IDs: IstanbulMU6
Record Dates: First submitted 2019-12-03; First posted 2019-12-20 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Psoriasis Vulgaris is a chronic, recurrent, inflammatory and hyperproliferative skin disease. Joint involvement is common along with skin involvement. However, metabolic diseases, such as cardiovascular diseases can be accompanied by many systemic diseases, chronic and repetitive due to the quality of life and psychological status of patients can affect. Today, although the treatment is repetitive, chronic and requires follow-up due to the disease patients can turn to alternative and complementary medicine techniques. In recent years, studies on alternative medicine and complementary therapies have been noted in the medical literature. These studies also include Case Reports related to psoriasis vulgaris. However, in our country, there is no study that tells us whether patients with psoriasis vulgaris apply these treatments or not and what the practitioners think about the success of the treatment. The aim of the study will be to clarify issues such as whether patients with Psoriasis Vulgaris apply alternative medicine and complementary therapies for their disease.

ELIGIBILITY:
Inclusion Criteria:

* psoriasis vulgaris patients

Exclusion Criteria:

* the patients that don't want to answer the questions

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: psoriasis vulgaris patients
Sampling Method: Non-Probability Sample
Enrollment: 1618 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Alternative medicine and complementary therapies that psoriasis vulgaris patients apply without informing the doctor, how they learn these techniques, what make them use these techniques for their illness | July 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Melek Aslan Kayıran, Istanbul, Turkey (Türkiye)